CLINICAL TRIAL: NCT03240757
Title: Metabolic Responses of a Single Bout of Low-intensity Exercise Following Mixed Meals in Healthy Individuals
Brief Title: Metabolic and Functional Impact of Various Breakfast Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Donato (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Livio Luzi, M.D., Full Professor of Endocrinology, Ospedale San Donato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Colazioni/1
Record Dates: First submitted 2017-08-01; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Metabolism and Nutrition Disorder
Keywords: meal absorption; exercise; energy balance; lipolysis
MeSH Terms: conditions — Nutrition Disorders; Motor Activity | interventions — Breakfast; Exercise

STUDY DESIGN:
Intervention Model Description: randomized-crossover in healthy subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breakfast without exercise (Active Comparator): Each subject of the same arm underwent 2 interventions: breakfast with/without exercise
  Interventions: Dietary Supplement: Breakfast
- Breakfast with exercise (Experimental): Each subject of the same arm underwent 2 interventions: breakfast with/without exercise
  Interventions: Dietary Supplement: Breakfast; Other: exercise

INTERVENTIONS:
Dietary Supplement: Breakfast — All subjects received a standard 75-g OGTT to assess eligibility for the study. The 19 subjects matching the inclusion criteria completed 2 experimental trials: resting and exercise. During the resting trial, all subjects underwent an OGTT (50-g: A) and 3 meal tolerance tests [one for each breakfast tested: B1 = milk (125ml) and cereals (30g); B2 = milk (220ml), apple (200g) and chocolate cream-filled sponge cake (30g); B3 = milk (125ml), apple (150g), bread (50g) and hazelnut chocolate cream (15g)]. In the exercise trial, 100 minutes after the glucose/meal ingestion, participants cycled for 20 min at 40% of maximum oxygen uptake.
Other: exercise — aerobic exercise at 40% of VO2max, for 20 minutes
  Arms: Breakfast with exercise

SUMMARY:
In the present study the investigators compared the hormonal and metabolic effects of three meal loads very popular among Italian eating habits, both in the resting- and exercising state. Given the lack of time is considered a common barrier to exercise adherence, we wanted to identify a low dose of exercise capable to produce health benefits in the post-absorptive status elicited by three commonly consumed meal-models in Mediterranean countries. To this end, healthy young volunteers firstly underwent an oral glucose tolerance test (OGTT) and three meal tolerance tests. Secondly, in an extra set of experiments, subjects cycled at low intensity for the last 20 minutes of the same glucose/meal tolerance test. Glycemia, insulinemia, ghrelinemia, lipidemia, and satiety were measured throughout OGTT and each test-meal load.

DETAILED DESCRIPTION:
The investigators evaluated postprandial responses (glucose, insulin, ghrelin, free fatty acids (FFA)) elicited by three diverse test-meal loads followed by a 20-min bout of low-intensity aerobic exercise were investigated. All subjects underwent a 50-g OGTT (A) and 3 test-meal loads: milk and cereals (B1); milk, apple and chocolate cream-filled sponge cake (B2); milk, bread, apple and hazelnut chocolate cream (B3). In the exercise trial, participants cycled for 20 minutes at 40% VO2max, 100 minutes after load ingestion.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 40 years
* normal body weight (BMI =18.5 - 24.9 according to NHLBI)
* stable diet

Exclusion Criteria:

* Diabetes, tipe 1 and 2 (ADA criteria)
* Glucose intolerance (ADA criteria)
* Dyslipidemia (ATP III according to NCEP)
* Metabolic syndrome

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2009-07-14 (Actual); Primary Completion 2010-05-28 (Actual); Study Completion 2010-05-28 (Actual)

PRIMARY OUTCOMES:
Plasma glucose responses of a single bout of low-intensity exercise following mixed meals in healthy individuals. | The entire study lasted for 9 experimental days (1 day for eligibility, 4 days for resting trial, 4 days for exercise trial).
  Postprandial glycemic responses elicited by three diverse test-meal loads followed by a 20-min bout of low-intensity aerobic exercise.
Plasma insulin responses of a single bout of low-intensity exercise following mixed meals in healthy individuals. | The entire study lasted for 9 experimental days (1 day for eligibility, 4 days for resting trial, 4 days for exercise trial).
  Postprandial insulinemic responses elicited by three diverse test-meal loads followed by a 20-min bout of low-intensity aerobic exercise.
Plasma ghrelin responses of a single bout of low-intensity exercise following mixed meals in healthy individuals. | The entire study lasted for 9 experimental days (1 day for eligibility, 4 days for resting trial, 4 days for exercise trial).
  Postprandial ghrelinemic responses elicited by three diverse test-meal loads followed by a 20-min bout of low-intensity aerobic exercise.
Plasma free fatty acids (FFA) responses of a single bout of low-intensity exercise following mixed meals in healthy individuals. | The entire study lasted for 9 experimental days (1 day for eligibility, 4 days for resting trial, 4 days for exercise trial).
  Postprandial plasma FFA responses elicited by three diverse test-meal loads followed by a 20-min bout of low-intensity aerobic exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Livio Luzi, M.D., Principal Investigator — Gruppo San Donato

IPD SHARING:
Plan to Share IPD: No
De-identified collective participant data for all outcome measures will be made available upon publication

REFERENCES:
- [Result] R Codella, A Caumo, S Benedini, M Adamo, A Ferrulli, C Macrì, I Terruzzi, L Luzi. Metabolic responses of a single bout of low-intensity exercise following mixed meals in healthy individuals. ADA (American Diabetes Association) 77th Scientific Session, 8-13 giugno 2017, San Diego, CA, USA. Diabetes 2017 Jun; 66 (Supplement 1).